CLINICAL TRIAL: NCT01638312
Title: The Development of Fast and Simple Method of Fructose Identification in Urine to Detect the Viral Infection in Early Stage
Brief Title: Development of Method of Fructose Identification in Urine to Detect the Viral Infection
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-20110188
Record Dates: First submitted 2012-01-20; First posted 2012-07-11 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV, fructose
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV infection patient and health people: The study does not have intervention

SUMMARY:
The goal of this research is the attempt to implement a new research method based on modern electrochemistry successes, in particular the development of the polarographic method of fructose and fructose diphosphate identification and its implementation to detect the viral infection in early stage. There will be 20 samples from the HIV-infected patients and 30 samples from the heath controls. The study will collect 10ml urine and examined fructose and fructose-diphosphate using the polarographic method.

DETAILED DESCRIPTION:
The goal of this research is the attempt to implement a new research method based on modern electrochemistry successes, in particular the development of the polarographic method of fructose and fructose diphosphate identification and its implementation to detect the viral infection in early stage.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection

Exclusion Criteria:

* who are in highly active antiretroviral therapy(HARRT) therapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the person who has HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JihJin Tsai, MD, Principal Investigator — The Medicines Company
Locations (1):
- Tropical Medicine Center, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- "HIV Infected Patients": The people had infected HIV
- "Healthy Controls": The people didn't have infected HIV
Period: Overall Study
Arm/Group | "HIV Infected Patients" | "Healthy Controls"
Started | 20 | 30
Completed | 20 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "HIV Infected Patients" | "Healthy Controls" | Total
Number analyzed (Participants) | 20 | 30 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 30 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.15 (10.27) | 31.87 (9.46) | 32.38 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 18 | 19
  Male | 19 | 12 | 31
Region of Enrollment [Number; unit: participants]
  Taiwan | 20 | 30 | 50

OUTCOME MEASURES:

1. Primary Outcome: Fructose Identification in Urine to Detect the Viral Infection : Number of Participants With Positive and Negative Waveform
Description: This detection technique, after a viral infection caused by the use of cell pathological changes and urine metabolic waste - fructose concentration, derivatives.Health News voltage changes to detect viral pathogens of activity and virulence. Because viral infection caused by the voltage change has its typical, So you can use voltage measurements to calibrate the presence and activity of a viral infection.
  1.How to interpretation the data The gap between values on X-axis is σ, and 50 is a reference to the center position. For example, the sample maybe contain with HIV virus if σ≧10 units.
  σ≧10 abnormal positive (+) σ<10 normal negative (-)
Time Frame: Participants provided urine samples once
Measure: Number; unit: participants
Groups:
- "HIV Infected Patients": 20 There are six medication negative response, referring to a recent comparison of the value of the blood virus date, there are three items detected waveform error, the remaining non-medication of 14, there are two detection waveform is negative; positive predictive value = 60%
- "Healthy Controls": Healthy people
  Graphical analysis of healthy people 1.7 of 30 healthy people were positive in waveform, and 23 were negative, the negative predictive value was 76.67%.
  2."Healthy people" was subjective judgments of participants, no other test as proof.
  3.Graphical analysis of HIV-infected subjects
Arm/Group | "HIV Infected Patients" | "Healthy Controls"
Number analyzed (Participants) | 20 | 30
participants
  Positive in waveform | 12 | 7
  Negative in waveform | 8 | 23

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected
Groups:
- "HIV Infected Patients"; "Healthy Controls": Serious and Other (Not Including Serious) Adverse Events were not collected
Arm/Group | "HIV Infected Patients" | "Healthy Controls"
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes